CLINICAL TRIAL: NCT00735423
Title: Effects of Neonatal Diet on Language, Neurocognitive Functions at Eight Years Old: fMRI, ERP and Standardized Behavioral Measures
Brief Title: Infant Diet Effects on Brain Function and Language Processing (fMRI)
Status: Active, not recruiting | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 77556
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Healthy
Keywords: Healthy children; Brain Function; Diet; Nutrition; Language; fMRI; ERP; Behavior
MeSH Terms: conditions — Language; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No groups: IDE used for outcome measurement not intervention
  Interventions: Device: No intervention

INTERVENTIONS:
Device: No intervention — IDE used for outcome measurement not intervention

SUMMARY:
The purpose of this study is to identify neurocognitive functions and language processing of 8-year-old children who were fed either breast milk, milk-based formula or soy-based formula during the first year of life.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 8-year-old children
* Full term
* Birth weight between the 5th - 95th weight-for-age
* Use of Breast milk, milk-based formula or soy-based formula throughout first year of life
* English as primary language
* Right handed first visit
* BMI between 5th - 95th percentile-for-age

Exclusion Criteria:

* Children with sleep disorders
* Children who use certain medications that may interfere with study assessments
* Illnesses or diseases or conditions that may interfere with study assessments

Ages: 90 Months to 101 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: healthy 8-year-old children
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Brain function test | 8 year old
Language processing tests | 8 year old

CONTACTS AND LOCATIONS:
Overall Officials: Xiawei Ou, Ph.D., Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Ou X, Andres A, Cleves MA, Pivik RT, Snow JH, Ding Z, Badger TM. Sex-specific association between infant diet and white matter integrity in 8-y-old children. Pediatr Res. 2014 Dec;76(6):535-43. doi: 10.1038/pr.2014.129. Epub 2014 Aug 28. PMID 25167204